CLINICAL TRIAL: NCT03825302
Title: Prostaglandin E2 as a Critical Mediator of Sex Disparities in Asthma
Status: Withdrawn | Type: Observational
Why Stopped: No funding available.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Cahill, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: PGE2 in asthma
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, blood, nasal fluid, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males with asthma: Induced sputum, methacholine challenge, and mannitol challenge will be performed.
  Interventions: Diagnostic Test: Methacholine challenge; Diagnostic Test: Mannitol challenge
- Females with asthma: Induced sputum, methacholine challenge, and mannitol challenge will be performed.
  Interventions: Diagnostic Test: Methacholine challenge; Diagnostic Test: Mannitol challenge

INTERVENTIONS:
Diagnostic Test: Methacholine challenge — Methacholine inhalation challenge will be administered to both male and females with asthma
Diagnostic Test: Mannitol challenge — Mannitol inhalation challenge will be administered to both male and females with asthma

SUMMARY:
This study seeks to understand how biological sex influences airway hyperresponsiveness in adult asthma.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and provide informed consent
* Age 18-50
* A history of physician-diagnosed asthma well controlled as assessed by ACQ-6 <1.5 and FEV1>70% of predicted and FEV1 >1.5 liters.
* Asthma must be persistent, defined by the requirement of a daily controller agent.
* Use of a stable dose of daily inhaled corticosteroids for the prior 3 months.
* Female subjects of childbearing potential must have a negative pregnancy test upon study entry and at each study visit.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* Hypogonadism, irregular menstrual cycles, polycystic ovarian syndrome (PCOS), exogenous hormonal supplements or contraception.
* Any chronic lung condition outside of asthma including chronic obstructive pulmonary disease (COPD), interstitial lung disease, eosinophilic granulomatosis with polyangiitis, allergic bronchopulmonary aspergillosis.
* Inability or unwillingness to hold the following medications prior to mannitol and methacholine inhalational challenge(s): Short-Acting Beta 2 Agonists >8 hours, Inhaled Corticosteroids and Anticholinergic Bronchodilators >12 hours, Phosphodiesterase Inhibitors or Adenosine Receptors >24 hours, Long-acting Beta 2 Agonists >36 hours, Long-acting Anticholinergics or Short-Acting Antihistamines >48 hours, Long-Acting Antihistamines >72 hours, and Leukotriene-Receptor Antagonist or 5-Lipooxygenase Inhibitors >4 days.
* For males, a screening morning serum total testosterone level (obtained between 8-10 AM) below the normal reference lab value.
* Current pregnancy, breast-feeding, or plans to become pregnant during the study period.
* Oral or systemic corticosteroid use or biologic agent for asthma in the previous 3 months or ED/Hospitalization for asthma within 6 months.
* Use of investigational drugs within 12 weeks of participation.
* Known hypersensitivity or allergy to mannitol, gelatin or methacholine.
* Upper or lower respiratory tract infection within the proceeding 6 weeks.
* A history of uncontrolled hypertension, coronary artery disease, stroke, epilepsy, urinary tract obstruction, untreated thyroid disease, or a chronic lung disease other than asthma.
* Daily use of a beta-blocker.
* Intolerance to anticholinergic medications.
* Inability to produce an adequate sputum sample.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Asthmatics at VUMC
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Provacative dose of mannitol that elicits a 15% decline in forced expiratory volume in males | Baseline
  Males only
Provacative dose of mannitol that elicits a 15% decline in forced expiratory volume in females | Baseline
  Females only during the luteal phase of the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Cahill, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided